CLINICAL TRIAL: NCT06071403
Title: The Effects of Time Points to Cease Parenteral Nutrition and IGF-1 on Very Low Birth Weight Infants--A Multicenter Prospective Cohort Study
Brief Title: The Effects of Time Points to Cease Parenteral Nutrition and IGF-1 on Very Low Birth Weight Infants
Status: Recruiting | Type: Observational
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Li Shuaijun, Postdoctor, Attending physician, Peking University
Other Study IDs: IRB00001052-23093
Record Dates: First submitted 2023-09-25; First posted 2023-10-06 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Growth Retardation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — The serum will be used to test the concentration of insulin-like growth factor 1.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- 60-70% group: We classified subjects into 3 groups by ((enteral feeding volume/total fluid volume)*100%).
  Interventions: Other: (enteral feeding volume/ total fluid volume)*100%
- 71-80% group: We classified subjects into 3 groups by ((enteral feeding volume/total fluid volume)*100%).
  Interventions: Other: (enteral feeding volume/ total fluid volume)*100%
- 81-90% group: We classified subjects into 3 groups by ((enteral feeding volume/total fluid volume)*100%).
  Interventions: Other: (enteral feeding volume/ total fluid volume)*100%

INTERVENTIONS:
Other: (enteral feeding volume/ total fluid volume)*100% — (enteral feeding volume/ total fluid volume)*100%. Total fluid volume is defined as enteral feeding volume + parenteral fluid volume + other fluid volume

SUMMARY:
This study aims to estimate short-term and long-term effects of time points to cease parenteral nutrition on very preterm infants, such as growth; to estimate the role of insulin-like growth factor 1 in the growth.

DETAILED DESCRIPTION:
At present, it is unclear when to cease parenteral nutrition, the effects of cessation times on preterm infants' growth, and whether insulin-like growth factor 1 (IGF-1) has a mediation effect in the procedure that nutrients regulate the growth in preterm infants.

Therefore, a prospective cohort study was designed with the aims:

1. to estimate the association between the time to cease parenteral nutrition and the growth in very low birth weight;
2. to investigate the relationship between nutrient volume in parenteral nutrition and growth in very low birth weight;
3. to analyze the IGF-1 mediation effect between nutrient volume and growth regulations.

ELIGIBILITY:
Inclusion Criteria:

1. Infants with a birth weight less than 1500 grams
2. Infants admitted within 72 hours after birth
3. Infants born from July 1, 2023, to June 30, 2024
4. Written informed consent from parents or guardians

Exclusion Criteria:

1. Infants with congenital abnormality
2. Infants surviving <7 days after birth

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Very low birth weight infants(birth weight less than 1500 grams)
Sampling Method: Non-Probability Sample
Enrollment: 416 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
short-term weight and long-term weight | at 36 weeks' corrected age (CA), CA 3 months, CA 6 months, CA 12 months, CA 18 months, CA 24 months, 36 months' age, 48 months' age and 60 months' age
  weight
short-term head circumference and long-term head circumference | at 36 weeks' corrected age (CA), CA 3 months, CA 6 months, CA 12 months, CA 18 months, CA 24 months, 36 months' age, 48 months' age and 60 months' age
  head circumference
short-term length and long-term length | at 36 weeks' corrected age (CA), CA 3 months, CA 6 months, CA 12 months, CA 18 months, CA 24 months, 36 months' age, 48 months' age and 60 months' age
  length

CONTACTS AND LOCATIONS:
Overall Officials: Shuaijun Li, doctor, Study Chair — Peking University
Locations (1):
- Wei Guo, Xingtai, Hebei, China